CLINICAL TRIAL: NCT00169897
Title: Effects of a Home-based Versus a Hospital-based Outpatient Pulmonary Rehabilitation Program in Patients With COPD: a Multicenter, Randomized Trial
Brief Title: Pulmonary Rehabilitation at Home Versus at the Gymnasium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Francois Maltais, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ISRCTN32824512
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2005-08

CONDITIONS: COPD
Keywords: COPD; Exercise; Self-management; Rehabilitation; Quality of life; Health economy; Cost effectiveness; Health care utilization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Patient Acceptance of Health Care | interventions — Educational Status; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital-based (Experimental): This group has to go at the hospital 3 times per week to do the exercise program.
  Interventions: Behavioral: Pulmonary rehabilitation (teaching and exercise)
- Home-Based (Active Comparator): The group had to do the exercise program at home with indirect supervision (Polar watches and a phone call per week).
  Interventions: Behavioral: Pulmonary rehabilitation (teaching and exercise)

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation (teaching and exercise) — After a 4-week education program, patients took part to home-based rehabilitation or outpatient hospital-based rehabilitation for 8 weeks. Patients were subsequently followed for 40 weeks to complete the one-year study.

SUMMARY:
Short term efficacy of pulmonary rehabilitation for improving functional capacity and quality of life of chronic obstructive respiratory disease (COPD) patient is well known. However, there is an important gap between the scientific knowledge and the clinical use of pulmonary rehabilitation since a a very small number of patients benefit from this therapeutic intervention. We estimate that less than 1% of the 750 000 canadians suffering from COPD have access to a pulmonary rehabilitation program. We want to study the efficacy of a home-based rehabilitation program as a way to facilitate the access to rehabilitation.

DETAILED DESCRIPTION:
This article on the main outcome is available. Maltais F, Bourbeau J, Shapiro S, Lacasse Y, Perrault H, Baltzan M, Hernandez P, Rouleau M, Julien M, Parenteau S, Paradis B, Levy RD, Camp P, Lecours R, Audet R, Hutton B, Penrod JR, Picard D, Bernard S. Effects of home-based pulmonary rehabilitation in patients with chronic obstructive pulmonary disease: a randomized trial. Ann Int Med 2008;149:869-878.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to ambulate. Defined as a 6MWD greater than 110 meters.
* Subject is diagnosed with COPD.
* 40 years-old and older
* Currently or previously smoking with a smoking history of at least 10 pack-years.
* Forced expiratory volume on one second (FEV1) after the use of a bronchodilator between 25 an 70% of the predicted value, and FEV1 to forced vital capacity ratio less than 70%.
* No previous diagnosis of asthma, left heart congestive heart failure (either radiographic evidence of pulmonary congestion, echocardiographic or ventriculographic evidence of a reduced ventricular ejection fraction), terminal disease, dementia or uncontrolled psychiatric illness.
* Never participated to a respiratory rehabilitation program and not staying or planning to stay in a long term care facility.
* Subject understands and is able to read and write French or English.
* MRC dyspnea scale of at least 2.

Exclusion Criteria:

* The need for supplemental oxygen at rest or during exercise will not be an exclusion criterion.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The dyspnea of the chronic respiratory questionnaire (CRQ) at 12 months is the primary outcome variable. | The data collection was terminated in January 2007 and publication was done December 2008
  Maltais F, Bourbeau J, Shapiro S, Lacasse Y, Perrault H, Baltzan M, Hernandez P, Rouleau M, Julien M, Parenteau S, Paradis B, Levy RD, Camp P, Lecours R, Audet R, Hutton B, Penrod JR, Picard D, Bernard S. Effects of home-based pulmonary rehabilitation in patients with chronic obstructive pulmonary disease: a randomized trial. Ann Int Med 2008;149:869-878.

SECONDARY OUTCOMES:
2-CRQ total score and specific domains, exercise tolerance (6MWD and submaximal exercise test) and ADL at 4 months. | The data collection was terminated in January 2007.
3-Health service utilization (physician and emergency department visits, hospitalizations) over the 1-year study period. | The data collection was terminated in January 2007.
4 Intervention cost. | The data collection was terminated in January 2007.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Maltais, MD, Principal Investigator — Laval University - Hopital Laval
Locations (10):
- Canada (10):
  - St-Paul's Hospital, Vancouver, British Columbia
  - Halifax Infirmary, Halifax, Nova Scotia
  - CRMSBC/Centre Hospitalier Baie-des-Chaleurs, Bonaventure, Quebec
  - Jewish Rehabilitation Hospital, Laval, Quebec
  - Hopital Hotel-Dieu de Levis, Lévis, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - Hopital Sacre-Coeur, Montreal, Quebec
  - Mount Sinai Hospital, Montreal, Quebec
  - CHA Enfant Jesus, Québec, Quebec
  - Hopital Laval, Sainte-Foy, Quebec

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Mak S, Bourbeau J, Mayo NE, Wood-Dauphinee S, Soicher JE. Psychometric Testing of the CHAMPS Questionnaire in French Canadians with COPD. Can Respir J. 2019 Sep 17;2019:2185207. doi: 10.1155/2019/2185207. eCollection 2019. PMID 31636770